CLINICAL TRIAL: NCT01412775
Title: The Contribution of a Short-term Psychological Group Intervention to Reduce Stress and Burnout Among Cardiac Intensive Care Nurses: A Pilot Study
Brief Title: Psychological Group Intervention to Reduce Stress and Burnout Among Cardiac Intensive Care Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MMC11XXX-XXCTIL
Record Dates: First submitted 2011-05-02; First posted 2011-08-09 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Stress, Psychological
Keywords: stress; burnout; exhaustion
MeSH Terms: conditions — Stress, Psychological; Burnout, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychological stress and exhaustion (Experimental): Twenty four male and female nurses from the cardiac intensive-care unit (CCU) of Meir Hospital, who consent to take part in the offered intervention program, will participate in the study. The participants will be randomly assigned to an experiment group of 12 participants and a control group of 12 participants.
  Interventions: Behavioral: short-term group intervention program

INTERVENTIONS:
Behavioral: short-term group intervention program — The intervention will include three aspects: Psycho-educational intervention: attending a lecture about stress and exhaustion; Techniques for decreasing stress: experiencing relaxation techniques and guided imagery and a BALINT style group:analyzing actual work cases and cognitive-behavioral focusing for reframing thoughts and making them more adaptive, expressing emotions and training for more appropriate behaviors.
  The study includes three weekly sessions, Each session will be 90 minutes in duration.
  Other Names: intervention program; short-term group intervention

SUMMARY:
The study will examine the influence of a Cognitive Behavioral Therapy (CBT) short-term group intervention program on the levels of psychological stress and professional exhaustion experienced by the nursing staff in a cardiac department.

DETAILED DESCRIPTION:
Exhaustion typifies a wide variety of professions, but it is especially evident in the service and aid professions (e.g., teaching and medicine), and nurses in particular are reported to be among the most exhausted. Exhaustion is described as nursing's "professional cancer", and stress is one of the major sources leading to it.

Articles and studies referring to stress among nurses in the years 1980-1996 mapped out six sources of stress stemming from inner sources related to the employee and those stemming from hospital organization: stress that stems from work patterns and overload (such as blurring, lack of clarity, lack of control and coping with death); interpersonal relationships at work (conflicts with other employees and with the medical staff); relationships with patients and their families (insufficient preparation for coping with the emotional needs of patients and their families); work organization and management (for example, lack of staff support and staff shortages); aspects related to the nursing profession (concerns regarding the treatment and care received by the patient), as well as concerns regarding the employee's practical knowledge and skills.

Since stress can lead, among other things, to functional exhaustion and dissatisfaction at work, and since studies have shown that stress has direct and indirect effects on the quality of patient care, it is important to find ways to decrease stress and the resulting exhaustion. Such efforts will increase nurses' efficiency at work and will also improve their quality of life, not to mention that of the patients. Therefore, the current study will examine the effectiveness of a short-term group intervention program for the nursing staff of a hospital's cardiac intensive-care unit.

There are a number of ways to decrease stress which vary both in the theory behind them ( the cognitive approach, for instance, explains the source of stress as stemming from cognitive and behavioral patterns acquired during one's life whereas the dynamic approach relates to deep and unconscious layers of the mind), and in their nature (the way in which they're facilitated). Researchers who have examined the relative efficacy of the different intervention programs in decreasing stress found that cognitive therapy is the most effective approach. Cognitive-behavioral therapy (CBT) can be applied both as individual therapy and as group therapy. According to the researchers, interventions in a group setting have several advantages over individual CBT: creating open relationships between staff members, giving participants an opportunity to get to know one another, providing a platform where employees can express their feelings, developing a sincere support group which proves crucial during stressful work situations, forging a feeling of belonging, and creative solving of shared conflicts and financial issues.

The current study will examine the influence of a CBT short-term group intervention program on the levels of psychological stress and professional exhaustion experienced by the nursing staff in a cardiac department.

The goal of the study:

The current study will examine the effectiveness of a short-term group intervention program for the nursing staff of a hospital's cardiac intensive-care unit. The intervention will include three aspects:

1. Psycho-educational intervention: attending a lecture about stress and exhaustion.
2. Techniques for decreasing stress: experiencing relaxation techniques and guided imagery.
3. A BALINT style group: analyzing actual work cases and cognitive-behavioral focusing for reframing thoughts and making them more adaptive, expressing emotions and training for more appropriate behaviors.

The study, which includes three weekly sessions, assumes that the intervention program will help to significantly decrease the participants' levels of psychological stress and professional exhaustion in comparison with their state before participation in the program, and also in comparison with those who didn't take part in the program (i.e., the control group).

The hypotheses of the study:

1. Participation in the intervention program will be related to decreased levels of psychological stress. The nursing staff in the program will demonstrate a lower level of negative psychological affect after participation. The level of stress will decrease significantly in comparison with the participants' state in the beginning of the program, and in comparison with professionals who didn't participate in the program (the control group).
2. Participation in the program will be related to reduced exhaustion levels: the nursing staff members who participate in the program will report lower exhaustion levels than they reported before the program, and in comparison with the control group (members of the nursing staff who didn't participate in the intervention program).

ELIGIBILITY:
Inclusion Criteria:

* Nurses from the cardiac intensive-care unit (CCU) of Meir Hospital, who consent to take part in the offered intervention program

Exclusion Criteria:

* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Symptoms of psychological stress | 6 weeks
  The Nursing Stress Scale (NSS) has been shown to be a valid and reliable instrument to assess occupational stressors among nurses.

SECONDARY OUTCOMES:
Exhaustion levels | 6 weeks
  Nurse's burnout symptoms: The SMBS questionnaire (Shirom-Melamed Burnout), will be used.This questionnaire reflects the participant's exhaustion in their workplace.

CONTACTS AND LOCATIONS:
Overall Officials: Morris Mosseri, Professor, Principal Investigator — Department of Cardiology, Meir Medical Center, Israel
Locations (1):
- Department of Cardiology, Meir Medical Center, Kfar Saba, Israel